CLINICAL TRIAL: NCT05472818
Title: SV2A Density Cannabis Use Disorder
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000032181; 1R01DA054314 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cannabis Use Disorder; Healthy
Keywords: Cannabis Use Disorder (CUD); Healthy subjects; synaptic vesicle density; [11C]APP311; UCB-J

STUDY DESIGN:
Intervention Model Description: In this study, patients with cannabis use disorder (CUD) and matched healthy controls will be scanned using anatomical magnetic resonance imaging (MRI) and PET. All participants will receive two PET scans, 4 weeks apart. CUD participants will be asked to abstain from cannabis for the 4 week period. A small subset of CUD participants will be asked to continue abstaining for an additional approx. 4 weeks to complete one additional scan. Participants may also complete a neurocognitive battery, various psychiatric evaluations, a physical examination, an ECG, blood tests, and questionnaires. CUD participants will complete bi-weekly study visits to confirm abstinence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CUD Group (Active Comparator): Participants will be scanned using anatomical magnetic resonance imaging (MRI) and PET. All participants will receive two PET scans, 4 weeks apart. CUD participants will be asked to abstain from cannabis for the 4 week period.
  Interventions: Drug: [11C]APP311
- Healthy Controls (Active Comparator): Participants will be scanned using anatomical magnetic resonance imaging (MRI) and PET. All participants will receive two PET scans, 4 weeks apart.
  Interventions: Drug: [11C]APP311

INTERVENTIONS:
Drug: [11C]APP311 — For each [11C]APP311 (UCB-J) PET scan, up to 20 mCi of [11C]APP311 (UCB-J) will be administered by infusion pump. All participants will receive at least two [11C]APP311 (UCB-J) PET scans approx. 4 weeks days apart. Approximately 8 CUD participants will be asked to return for a third [11C]APP311 (UCB-J) PET scan after an additional 4 weeks following their second scan.

SUMMARY:
The main purpose of this study is to determine whether hippocampal synaptic vesicle density estimated by hippocampal [11C]APP-311/[11C]UCB-J binding in individuals diagnosed with cannabis use disorder (CUDs) improves with at least 4 weeks of confirmed abstinence from cannabis, in comparison to healthy controls (HCs). Furthermore, any change in synaptic vesicle density will be placed in functional context by measuring verbal memory, which is sensitive to hippocampal function, before and after at least 4 weeks of confirmed abstinence. Finally, the relationship between hippocampal [11C]UCB-J binding in CUDs with measures of cannabis exposure (e.g., age of initiation, cumulative lifetime dose) will be explored.

ELIGIBILITY:
CUD Participants Inclusion Criteria:

1. Able to provide informed consent
2. Male and female 18-75 years old
3. Daily cannabis use
4. Positive urine screen for cannabinoids and negative for all other drugs on
5. Diagnosis of DSM-5 cannabis use disorder (≥ moderate, i.e., ≥ 4 [of 11] symptoms).
6. Must express a willingness at screening to set a date to attempt to quit using cannabis.
7. Physically healthy i.e., no clinically unstable medical conditions.
8. For women of childbearing potential (WOCBP) and men, willingness to practice birth control and to inform study staff immediately if either they (for women) or their partner (for men) becomes pregnant.
9. Additional criteria not disclosed here in order to minimize the risk of ineligible subjects enrolling in the study.

CUD Participants Exclusion Criteria:

1. Laboratory tests with clinically significant abnormalities or positive urine toxicology screen with exception of cannabinoids.
2. Women with a positive pregnancy test or women who are lactating.
3. Have implanted or embedded metal objects or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field
4. Have had exposure to ionizing radiation that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits.
5. History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto) Subjects who have donated blood within 8 weeks of the present study
6. Medications that could alter synaptic density and, therefore, confound the interpretation of study data.
7. Additional criteria not disclosed here in order to minimize the risk of ineligible subjects enrolling in the study.

Healthy Controls Inclusion Criteria:

1. Willing and able to give voluntary written informed consent
2. Male and Female subjects, age 18 to 75 years, inclusive
3. BMI within 19 to 35 kg/m2, inclusive
4. Must be in good health as determined by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests.
5. Negative urine drug screen
6. If female, not pregnant or breastfeeding
7. If female of childbearing potential, must agree to use an acceptable method of birth control, as determined by the principal investigator, for the duration of the study and up to one month after completion of PET scans.
8. Able to read and write, able to communicate effectively with the investigator, and comply with all study requirements, restrictions, and directions of the clinic staff.
9. Have arterial access sufficient to allow blood sampling as per the protocol.

Healthy Controls Exclusion Criteria:

1. History or presence of clinically significant and unstable respiratory, GI, renal, hepatic, pancreatic, hematological, neurological (including history of seizure), cardiovascular, psychiatric (including known addictive disorders), musculoskeletal, genitourinary, immunological, or dermatological disorders, including all cancers.
2. Abnormal clinically significant laboratory or physical findings during screening
3. History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto)
4. A condition that, in the opinion of the investigator, would prevent compliance with the study protocol.
5. Medications that could alter synaptic density and, therefore, confound the interpretation of study data.
6. MRI incompatible implants and other contraindications for MRI, such as pace-maker, artificial joints, non-removable body piercings, metal fragments in head and/or body, or history working with ferrous metals either as a vocation or hobby in such a way that might have led to unknown, indwelling metal fragments that could cause injury during MRI etc.
7. Subjects who suffer from claustrophobia.
8. Participation in other research studies involving ionizing radiation within one year of the PET scans that would cause the subject to exceed the yearly dose limits for healthy volunteers
9. Additional criteria not disclosed here in order to minimize the risk of ineligible subjects enrolling in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Hippocampal SV2A synaptic density | All participants will receive at least two [11C]APP311 (UCB-J) PET scans approx. 4 weeks days apart.
  Hippocampal SV2A synaptic density will be measured using [11C]APP311 (UCB-J).

SECONDARY OUTCOMES:
Hippocampal binding and Hippocampal Verbal Memory Task | The Auditory Verbal Learning Task (AVLT) will be administered before and after the 4 week abstinence period.
  To determine the relationship between hippocampal [11C]APP311 (UCB-J) binding and performance on the hippocampal verbal memory task (Auditory Verbal Learning Task [AVLT]), a cognitive task that measures total immediate recall, before and after 4 weeks of confirmed cannabis abstinence.
Hippocampal binding and Groton Maze Learning in CUDs | The Groton Maze Learning Task will be administered before and after the 4 week abstinence period.
  To determine the relationship between hippocampal [11C]APP311 (UCB-J) binding and performance on the Groton Maze Learning task, a cognitive task that measures total number of errors, in CUDs before and after 4 weeks of confirmed cannabis abstinence.

OTHER OUTCOMES:
Hippocampal synaptic density and first age of cannabis exposure | Before and after the 4 week abstinence period.
  To determine the relationship between hippocampal synaptic density (n=26+12 historical data) and indices of cannabis exposure such as first age of cannabis exposure, as measured by self-report data.
Hippocampal synaptic density and cumulative lifetime cannabis exposure. | Before and after the 4 week abstinence period.
  To determine the relationship between hippocampal synaptic density (n=26+12 historical data) and indices of cannabis exposure such as cumulative lifetime cannabis exposure, as measured by self-report data.
Hippocampal SV2A synaptic density after 8 weeks | Approximately 8 CUD participants will be asked to return for a third [11C]APP311 (UCB-J) PET scan after an additional 4 weeks following their second scan. (8 weeks in total).
  To explore whether hippocampal synaptic density and function continues to improve with 8 weeks of abstinence in a subset of CUD participants using [11C]APP311 (UCB-J).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States